CLINICAL TRIAL: NCT00125216
Title: Evaluation of the Effects of Response Elaboration Training for Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C3719-R
Record Dates: First submitted 2005-07-27; First posted 2005-07-29 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Aphasia; Language Disorders; Speech Disorders
Keywords: Aphasia; Language Therapy; Rehabilitation of speech and language disorders; Speech-language pathology
MeSH Terms: conditions — Aphasia; Language Disorders; Speech Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other): Single subject design - participant receives three administrations of the same treatment
  Interventions: Behavioral: Response Elaboration Training

INTERVENTIONS:
Behavioral: Response Elaboration Training — Therapist modeling, reinforcement and forward-chaining are used to stimulate verbal descriptions of pictures

SUMMARY:
The purpose of this study is to evaluate the effects of Response Elaboration Training (RET), which is a speech/language therapy for aphasia. The study is designed to determine whether verbal language production improves in terms of content and length of utterances as a result of treatment.

DETAILED DESCRIPTION:
Detailed Description:

Extended description of the protocol, including information not already contained in other fields, such as comparison(s) studied.

Example:

Sudden out-of-hospital cardiac arrest (OOH-CA) remains a significant cause of death, in spite of recent declines in overall mortality from cardiovascular disease. Existing methods of emergency resuscitation are inadequate due to time delays inherent in the transport of a trained responder with defibrillation capabilities to the side of the OOH-CA victim. Existing Emergency Medical Services (EMS) systems typically combine paramedic Emergency Medical Technician (EMT) services with some level of community involvement, such as bystander cardiopulmonary resuscitation (CPR) training. Some communities include automated external defibrillators (AEDs) at isolated sites or in mobile police or fire vehicles. A comprehensive, integrated community approach to treatment with AEDs would have community units served by these volunteer non-medical responders who can quickly identify and treat a patient with OOH-CA. Such an approach is termed Public Access Defibrillation (PAD).

Comparison(s): Community units trained and equipped to provide public access defibrillation in addition to optimal standard care, compared to community units trained to provide optimal standard care (recognition of out-of-hospital cardiac arrest, 911 access, and cardiopulmonary resuscitation).

The purpose of the proposed research is to thoroughly evaluate the effects of Response Elaboration Training (RET) with persons with aphasia. Specifically, the proposed research investigation is designed to delineate the outcomes that may be expected with RET. The study is also designed to improve outcomes in the area of stimulus generalization effects of treatment by testing a modification of RET designed to facilitate generalization. The specific experimental questions to be addressed are as follows:

* Will RET result in increased production of correct information units and increased length and changes in composition of utterances as measured in *trained and untrained picture descriptions; *story retells; *conversations with significant others/family members/friends; and *personal recounts?
* Will modification and extension of RET to additional training contexts result in further increases in production of CIUs and increased length and complexity of utterances?
* Will the effects* of RET vary among participants with fluent aphasia, participants with nonfluent aphasia who present with mild to moderate verbal production deficits, and participants with nonfluent aphasia who present with severe verbal production deficits?

  * Effects = effects on production of CIUs and on measures of functional communication
* Will changes in measures of functional communication be observed following administration of RET?

A series of single-subject experimental designs across subjects, behaviors, and contexts will be conducted to address these questions. Twenty-four adults with chronic, moderate to severe aphasia secondary to unilateral, left-hemisphere brain-injury will serve as participants for this investigation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe nonfluent or fluent aphasia
* Nonverbal intelligence within normal limits
* Auditory and visual acuity adequate for experimental tasks
* 6 months post-onset of single, focal brain injury (e.g., stroke)

Exclusion Criteria:

* Previous history of therapy with RET
* Diagnosed psychological disorder other than depression
* Neurological condition other than that which resulted in aphasia
* History of alcohol or substance abuse
* Non-native English speaker
* Premorbid history of speech/language disorder

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2004-12; Primary Completion 2007-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
verbal production of meaningful content words in connected speech | 3 and 6 weeks following completion of treatment
  Participants were asked to describe pictured scenes and to provide a monologue on a topic of their choice. Their speech/language was audio recorded during these tasks and recordings were transcribed by project speech/language pathologists. Counts of content words were made.

CONTACTS AND LOCATIONS:
Overall Officials: Julie L. Wambaugh, PhD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, Salt Lake City, Utah, United States

REFERENCES:
- [Result] Wambaugh JL, Nessler C, Wright S. Modified response elaboration training: application to procedural discourse and personal recounts. Am J Speech Lang Pathol. 2013 May;22(2):S409-25. doi: 10.1044/1058-0360(2013/12-0063). PMID 23695913